CLINICAL TRIAL: NCT06234059
Title: Behavioral and Neural Measures of Speech Motor Control
Brief Title: Modulation of Sensory Acuity With Transcranial Magnetic Stimulation (TMS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Another research group ran a similar study and reported results
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-1128 TMS (Exp 8); 1R01DC019134-01A1 (NIH); Protocol Version 4/29/2025 (Other: UW Madison); A481800 (Other: UW Madison)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-09

CONDITIONS: Speech
Keywords: speech motor control; vocal learning
MeSH Terms: conditions — Speech | interventions — Transcranial Magnetic Stimulation; Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adult Speakers (Experimental): healthy adult participants across the lifespan in three groups:18-35, 36-55, and 56+
  Interventions: Device: TMS; Behavioral: Speaking Tasks

INTERVENTIONS:
Device: TMS — This paradigm uses theta-burst transcranial magnetic stimulation (tbTMS) to modulate the excitability of sensory cortices to examine the effect on sensory acuity and sensorimotor adaptation. Participants will complete three total sessions targeting primary somatosensory cortex (S1): one using intermittent theta-burst stimulation (iTBS), one using continuous theta-burst stimulation (cTBS), and one with sham stimulation.
  Other Names: transcranial magnetic stimulation (continuous and intermittent theta-burst stimulation), electromyography (EMG)
Behavioral: Speaking Tasks — Participants will produce four training words under a vowel centralization feedback paradigm in which auditory feedback is altered. The investigators will measure changes in produced vowels as a result of the altered feedback in concert with the different stimulation regimes described in the TMS intervention.

SUMMARY:
The purpose of this research study is to understand how the brain processes and controls speech in healthy people. The investigators are doing this research because it will help identify the mechanisms that allow people to perceive their own speech errors and to learn new speech sounds, which may be applied to people who have communication disorders. 15 participants will be enrolled into this part of the study and can expect to be on study for 4 visits of 2-4 hours each.

DETAILED DESCRIPTION:
The overall study (Establishing the clinical utility of sensorimotor adaptation for speech rehabilitation) aims to understand how cognitive, perceptual, and motor processes are integrated in the control of speech movements. The investigators study how this complex skill is performed in healthy speakers to understand how this system functions, how this skill relates to the perception of speech, and what role different parts of the brain play in this process. Different studies look at how speech motor control is executed, maintained, and changed. Overall, the study will recruit 329 participants over the course of 5 years. Participants can expect to be on study for up to 3 weeks.

The entire study is composed of 8 experiments and 6 interventions. The present record represents the experiments involving transcranial magnetic stimulation (TMS), i.e. Experiment 8: Modulating sensorimotor adaptation through TMS to somatosensory cortex.

This paradigm uses theta-burst transcranial magnetic stimulation (tbTMS) to modulate the excitability of sensory cortices to examine the effect on sensory acuity and sensorimotor adaptation. Participants will complete three total sessions targeting primary somatosensory cortex (S1): one using intermittent theta-burst stimulation (iTBS), one using continuous theta-burst stimulation (cTBS), and one with sham stimulation.

The effect of the stimulation on somatosensory adaptation will be measured using a vowel centralization feedback perturbation experiment: after stimulation, participants will produce words under conditions of altered auditory feedback, and the investigators will measure changes in produced vowels as a result of these alterations.

ELIGIBILITY:
Inclusion Criteria (Control):

* English-speaking adults
* normal hearing and speech
* no history of stroke or neurological conditions

Exclusion Criteria:

* Native language other than English
* Any neurological disorders other than the disorder of interest
* Any history of hearing disorders
* Uncorrected vision problems that prevent participants from seeing visually-presented stimuli
* Significant cognitive impairments that prevent participants from carrying out the task or from giving informed consent
* Vulnerable populations (minors and prisoners)
* Additional exclusionary criteria for TMS:

  * Implanted paramagnetic materials (metal clips, plates, pacemakers, etc.)
  * Increased risk in the event of a seizure
  * Serious heart disease
  * Increased intracranial pressure
  * Pregnancy
  * History of seizures
  * Family history of epilepsy
  * Epileptogenic medications
  * Chronic or transient disruption of sleep (including jet lag)
  * History of fainting
  * Chronic or transient increase in stressful experiences
  * Use of illegal drugs
  * If the TMS visit involves a visual acuity task at the same time as TMS] Use of glasses at the research study visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Acoustic vowel space measures: AVS (acoustic vowel spacing)/VSA (vowel space area) | up to 1 hour
  For speech production tasks, the primary acoustic measure will be adaptation to the altered feedback, defined here as increases in AVS (average vowel spacing), the mean of pairwise formant distances between vowels. The investigators will also include a global measure of working vowel space, the quadrilateral vowel space area (qVSA). qVSA measures the area (in Hz^2) between the F1/F2 coordinates of the corner vowels. Both the more local AVS and more global qVSA have been linked to speech intelligibility in various types of dysarthria.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Niziolek, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Link to study record for experiment 7 [NCT05723575] — https://clinicaltrials.gov/study/NCT05723575
- See also: Link to study record for experiment 5 [NCT05286658] — https://clinicaltrials.gov/study/NCT05286658